CLINICAL TRIAL: NCT06416397
Title: Diagnostic Approach for Cholangiocarcinoma Using Liquid Bile Biopsy
Acronym: PROTEOBILE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/69
Record Dates: First submitted 2024-02-01; First posted 2024-05-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Diagnosis; Cancer; Proteomic profiling
MeSH Terms: conditions — Cholangiocarcinoma; Disease; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Proteomic profile — Proteomic analysis of bile samples will be performed every 5 bile samples. Bile samples will be taken during endoscopy with retrograde papillary catheterization or radiological procedures in selected patients. In clinical practice, bile samples are taken for bacteriological purposes. An average of 10 mL is taken.
  Five mL are required for bacteriological analysis. The remaining millilitres, which are usually discarded, will be kept for storage and to form the bile bank at the Biological Resources Centre before to be analyzed in proteomics.

SUMMARY:
The main aim of the study is to develop a diagnostic proteomic profile of cholangiocarcinoma using bile samples. The primary endpoint will be the rate of concordant positive diagnoses obtained from bile samples based on proteomic profiling compared with histological reference diagnoses (concomitant cytological sampling and/or final histological sampling).

DETAILED DESCRIPTION:
Cholangiocarcinoma has a poor 5-year prognosis (less than 5%) and is rarely resectable at diagnosis. Diagnosis is made by histological sampling (biopsy or endo-biliary brushing) during endoscopic retrograde catheterization of the papilla or radiologically during transparietohepatic drainage. Conventional histology techniques have a low sensitivity of around 14-60%, which leads to diagnostic delays, repeated invasive examinations and delays in therapeutic management, sometimes with progression from a resectable to an unresectable stage.

New techniques are emerging to optimize the diagnosis of cholangiocarcinoma, in particular molecular techniques. This is the case with proteomics and proteomic profiling, which consists of obtaining diagnostic information from all the proteins contained in biological samples.

Furthermore, during diagnostic procedures for cholangiocarcinoma, bile samples are taken, initially for bacteriological purposes. Proteomics has been shown to be a tool capable of identifying potential diagnostic biomarkers in bile samples. To date, proteomic profiling has never been tested on bile samples for diagnostic purposes, although its proof of concept has been established.

Obtaining a proteomic profile for the diagnosis of cholangiocarcinoma from bile samples would enable the development of an innovative tool that has not yet been described in this field. It would optimize the management of patients with cholangiocarcinoma, with the possibility of a quicker diagnosis enabling optimal management as soon as the first clinical symptoms appear, while reducing the number of examinations required to obtain a diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years and older
* Patients with bile duct stenosis who require endoscopy with retrograde papillary catheterization or a radiological procedure for diagnostic purposes (histological samples) as part of their management
* Oral consent

Exclusion Criteria:

* Pregnant woman
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with bile duct stenosis who require ERCP or a radiological procedure for diagnostic purposes (histological samples) as part of their management
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
positive diagnosis of cholangiocarcinoma | Baseline
  rate of positive diagnosis of cholangiocarcinoma obtained from bile samples using proteomic profile analysis compared with the rate of positive diagnosis using histological reference tools.

SECONDARY OUTCOMES:
Identification of diagnostic biomarkers for cholangiocarcinoma | Baseline
  pecific analysis of proteomic data to identify a recurrent, malignancy-specific target protein
differential diagnosis rates | Baseline
  differential diagnosis rates obtained by proteomic profiling compared with histological results
positive diagnoses with the Next-Generation Sequencing technique | Baseline
  rate of positive diagnoses with the Next-Generation Sequencing technique

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No